CLINICAL TRIAL: NCT03761693
Title: Fasting Tolerance in Patients With Medium-chain Acyl-CoA Dehydrogenase Deficiency (MCADD) in the First Six Months of Life: an Investigator-initiated Human Pilot-study
Brief Title: Fasting Tolerance in MCADD-infants
Acronym: FiTtINg MCADD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Terry G.J. Derks, MD, PhD, Principal Investigator, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL201800774
Record Dates: First submitted 2018-11-21; First posted 2018-12-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Mcad Deficiency
Keywords: Mcad deficiency; Phenotypic Variation; Biomarkers; Diet Therapy
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe/classical MCADD (Experimental): Severe MCADD will be defined by ACADM mutations associated with clinical ascertainment or residual MCAD enzyme activity < 10 %, as defined previously (Touw et al., 2012).
  Interventions include fasting challenges at two and six months of age.
  Interventions: Other: Fasting test
- Mild MCADD (Experimental): Mild MCADD will be defined by the remaining ACADM genotype variants and residual MCAD enzyme activity ≥ 10%.
  Interventions include fasting challenges at two and six months of age.
  Interventions: Other: Fasting test

INTERVENTIONS:
Other: Fasting test — The included infants will be fasted according to local standardized procedures at the University Medical Centre Groningen. Fasting will take place under hourly blood glucose monitoring and bedside supervision by an experienced, dedicated pediatric nurse, in collaboration with a metabolic pediatrician, who will be available to attend the patient instantly. Furthermore, on request of parent(s) or guardian(s), a continuous blood glucose monitoring device can be used during the study visits.
  During study visit 1, at two months of life, fasting will be continued for maximally eight hours.
  During study visit 2, at six months of life, fasting will be continued for maximally twelve hours.
  Fasting will be ended prematurely in the following events:
  * blood glucose concentration drops < 3.6 mmol/L;
  * the child shows symptoms/signs of a low blood glucose concentration;
  * patients parent(s) or guardian(s) request end of fast.

SUMMARY:
MCAD deficiency (MCADD; #OMIM 201450) is the most common inherited disorder of mitochondrial fatty acid oxidation. Already before the introduction of population newborn bloodspot screening (NBS), large phenotypic heterogeneity was observed between MCADD-patients, ranging between deceased patients and asymptomatic subjects. Most clinically ascertained patients were homozygous for the common c.985A>G ACADM mutation. After NBS, newborns with novel ACADM-genotypes have been identified and subjects can be classified as either severe/classical or mild/variant MCADD-patients.

Dietary management guidelines are based on expert opinion, limited experimental data summarized in one retrospective study on fasting tolerance in 35 MCADD patients. Interestingly, data are absent from fasting tolerance in MCADD patients between 0-6 months of age. These guidelines cause parental stress, especially for young patients. Moreover, the guidelines do not take into account the heterogeneity between patients, including the classification between severe versus mild MCADD-patients. The investigators question whether at least a subset of the MCADD-patients is overtreated with these guidelines.

Therefore, the investigators propose this pilot-study on fasting tolerance in 10 subjects with severe MCADD and 10 subjects with mild MCADD at the ages of two and six months. Differences between subsets of MCADD-patients will be studied longitudinally by both traditional metabolic parameters and unbiassed metabolomics, lipidomics and proteomics approach. This project will substantiate current management guidelines and aims to identify new (prognostic) biomarkers.

DETAILED DESCRIPTION:
Rationale: MCAD deficiency (MCADD; #OMIM 201450) is the most common inborn error of mitochondrial fatty acid oxidation. Already before the introduction of population newborn bloodspot screening (NBS), large phenotypic heterogeneity was observed between MCADD patients, ranging between deceased patients and asymptomatic subjects. Most clinically ascertained patients were homozygous for the common c.985A>G ACADM mutation. After the introduction of the disorder to the NBS, newborns with novel ACADM-genotypes have been identified. Subjects can be classified as either severe/classical or mild/variant MCADD patients. Dietary management guidelines are based on expert opinion and limited experimental data summarized in one retrospective study on fasting tolerance in 35 MCADD-patients. Interestingly, data are absent from the fasting tolerance of MCADD patients between 0-6 months of age. These guidelines cause parental stress, especially regarding young patients (0-6 months). Moreover, the guidelines do not take into account the heterogeneity between patients, including the classification between severe versus mild MCADD patients. The investigators question whether at least a subset of the MCADD patients is overtreated with these guidelines.

Objective: The main objective of the study is to explore the fasting tolerance in MCADD-patients of two and six months of life. Second, it is aimed to compare fasting tolerance and biochemical dynamics between subsets of MCADD patients. Third, it is aimed to identify novel diagnostic and/or prognostic biomarkers. The last objective is to elucidate the (fundamental) origin of phenotypical differences between MCADD patients.

Study design: Longitudinal, prospective investigator-initiated human pilot-study.

Study population: Otherwise healthy infants with severe MCADD and mild MCADD at the ages of two and six months of life.

Intervention: During two visits, the included infants will be fasted according to local standardized procedures at the University Medical Centre Groningen (UMCG). Fasting will take place under continuous blood glucose monitoring and bedside supervision by an experienced, dedicated pediatric nurse in collaboration with a metabolic pediatrician, who will be available to attend the patient instantly. During visit 1, at two months of life, fasting will be continued for maximally eight hours. During visit 2, at six months of life, fasting will be continued for maximally twelve hours. Fasting will be ended prematurely if; (a) the blood glucose concentration drops < 3.6 mmol/L, (b) the fasting subject shows symptoms/signs of a low blood glucose concentration, and/or (c) subject's parent(s) or guardian(s) request the end of fast.

Main study parameters/endpoints: Dynamics of both traditional clinical and biochemical metabolic parameters and unbiased multi-omics (metabolomics, lipidomics, and proteomics) parameters will be studied.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The trial is considered to be a low-risk study. The clinical research team at the UMCG has a longstanding tradition of performing supervised controlled clinical fasting test in patients with inborn errors of metabolism, for diagnostic as well as research purposes. No adverse effects are expected during fasting in otherwise healthy infants with MCADD. The study holds three moderate burdens for participants: insertion of the indwelling IV catheter, the discomfort of fasting for the subject and the parent(s) or guardian(s), and the time consumption. However, subjects and their parents(s) may directly benefit from the results of this study by reduction of stress concerning feeding, under normal, healthy circumstances and the (possible) institution of a personalized feeding regimen based on the study results by the treating pediatrician. As this project will substantiate current management guidelines and aims to identify new (prognostic) biomarkers, it may further improve the outcomes of future MCADD patients and their parent(s) or guardian(s), by reduction of (unnecessary) parental stress, treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* A child must be at least younger than 6 months of life at inclusion. In case of prematurity, the child will be included and treated according to the adjusted age.
* Established MCADD diagnosis. The diagnosis should be confirmed by a combination of (a) NBS outcome (b) MCAD enzyme activity measured with phenylpropionyl-CoA as a substrate, ideally in lymphocytes (considered to be the golden standard) and (c) ACADM gene mutation-analysis.

Exclusion Criteria:

* Any other chronic and/or genetic condition that is deemed an exclusion criterion based on the judgement of the treating metabolic paediatrician.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose concentrations | Up to 8 samples will be taken during the maximally 8 hour fast (session 1), up to 12 samples will be taken during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (8:00 AM) and hereafter hourly during the fast of session 1 and session 2.
Change in plasma free fatty acid (FFA) concentrations | Up to 8 samples will be taken during the maximally 8 hour fast (session 1), up to 12 samples will be taken during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (8:00 AM) and here-after hourly during the fast of session 1 and session 2.
Change in Heart rate | Up to 8 frequencies will be noted during the maximally 8 hour fast (session 1), up to 12 frequencies will be noted during the maximally 12 hour fast (session 2)
  Heart rate per minute will be noted at baseline (8:00 AM) and here-after hourly during the fast of session 1 and session 2.
Change in Respiratory rate | Up to 8 frequencies will be noted during the maximally 8 hour fast (session 1), up to 12 frequencies will be noted during the maximally 12 hour fast (session 2).
  Respiratory rate per minute will be noted at baseline (8:00 AM) and here-after hourly during the fast of session 1 and session 2.
(Change in) presence of lethargy | Up to 8 physical examinations will be performed during the maximally 8 hour fast (session 1), up to 12 physical examinations will be performed during the maximally 12 hour fast (session 2). Physical examinations will take 5 minutes.
  Physical examination will be performed hourly by a nurse during the fast of session 1 and session 2.
  Yes/no; if yes, #hours, minutes.
(Change in) presence of trembling | Up to 8 physical examinations will be performed during the maximally 8 hour fast (session 1), up to 12 physical examinations will be performed during the maximally 12 hour fast (session 2). Physical examinations will take 5 minutes.
  Physical examination will be performed hourly by a nurse during the fast of session 1 and session 2.
  Yes/no; if yes, #hours, minutes.

SECONDARY OUTCOMES:
Continuous glucose monitoring (CGM) data | Blood glucose concentrations will be sensored every 5 minutes, during the maximally 8 hour fast (session 1). Blood glucose concentrations will be sensored every 5 minutes, during the 12 hour fast (session 2).
  Subcutaneous glucose concentrations will be obtained with a Dexcom G6 CGM sensor, if used.
Blood pH | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Blood oxygen partial pressure | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Blood carbon dioxide partial pressure | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Plasma bicarbonate concentrations | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Base excess | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Blood oxygen saturation | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Plasma ketones concentrations (β-hydroxybutyrate, acetoacetate) | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (hours, minutes).
Plasma acylcarnitines concentrations | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (hours, minutes).
Plasma amino acid concentrations | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Urine organic acids concentrations | 2 samples will be collected during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  During session 1, sample #1 will be collected during the first 6 hours of the maximally 8 hours fast. Sample #2 will be collected during the last 2 hours of the maximally 8 hour fast. During session 2, sample #1 will be collected during the first 10 hours of the maximally 12 hour fast. Sample 2 will be collected during the last 2 hours of the maximally 12 hour fast.
(Untargeted) Metabolomics | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Lipidomics | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the maximally 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).
Proteomics | 3 samples will be taken during the maximally 8 hour fast (session 1) and during the 12 hour fast (session 2).
  Sample #1 will be collected at baseline (start fast, 8:00 AM), sample #2 will be collected 2 hours after the start of the fast (10:00 AM), sample #3 will be taken at the end of the fast after maximally 8 hours (16:00, session 1) or 12 hours (20:00, session 2), or earlier if necessary (#hours, minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Terry Derks, MD, PhD, Principal Investigator — Consultant pediatrician metabolic diseases
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derks TG, van Spronsen FJ, Rake JP, van der Hilst CS, Span MM, Smit GP. Safe and unsafe duration of fasting for children with MCAD deficiency. Eur J Pediatr. 2007 Jan;166(1):5-11. doi: 10.1007/s00431-006-0186-0. Epub 2006 Jun 21. PMID 16788829
- [Background] Touw CM, Smit GP, de Vries M, de Klerk JB, Bosch AM, Visser G, Mulder MF, Rubio-Gozalbo ME, Elvers B, Niezen-Koning KE, Wanders RJ, Waterham HR, Reijngoud DJ, Derks TG. Risk stratification by residual enzyme activity after newborn screening for medium-chain acyl-CoA dehyrogenase deficiency: data from a cohort study. Orphanet J Rare Dis. 2012 May 25;7:30. doi: 10.1186/1750-1172-7-30. PMID 22630369
- [Background] Fletcher JM, Pitt JJ. Fasting medium chain acyl-coenzyme A dehydrogenase--deficient children can make ketones. Metabolism. 2001 Feb;50(2):161-5. doi: 10.1053/meta.2001.20177. PMID 11229423
- [Background] Heales SJ, Thompson GN, Massoud AF, Rahman S, Halliday D, Leonard JV. Production and disposal of medium-chain fatty acids in children with medium-chain acyl-CoA dehydrogenase deficiency. J Inherit Metab Dis. 1994;17(1):74-80. doi: 10.1007/BF00735398. PMID 8051939
- [Background] Jakobs C, Kneer J, Martin D, Boulloche J, Brivet M, Poll-The BT, Saudubray JM. In vivo stable isotope studies in three patients affected with mitochondrial fatty acid oxidation disorders: limited diagnostic use of 1-13C fatty acid breath test using bolus technique. Eur J Pediatr. 1997 Aug;156 Suppl 1:S78-82. PMID 9266222
- [Background] Walter JH. Tolerance to fast: rational and practical evaluation in children with hypoketonaemia. J Inherit Metab Dis. 2009 Apr;32(2):214-7. doi: 10.1007/s10545-009-1087-y. Epub 2009 Mar 4. PMID 19255872
- [Background] Bonnefont JP, Specola NB, Vassault A, Lombes A, Ogier H, de Klerk JB, Munnich A, Coude M, Paturneau-Jouas M, Saudubray JM. The fasting test in paediatrics: application to the diagnosis of pathological hypo- and hyperketotic states. Eur J Pediatr. 1990 Dec;150(2):80-5. doi: 10.1007/BF02072043. PMID 2279514
- [Background] Derks TG, Duran M, Waterham HR, Reijngoud DJ, Ten Kate LP, Smit GP. The difference between observed and expected prevalence of MCAD deficiency in The Netherlands: a genetic epidemiological study. Eur J Hum Genet. 2005 Aug;13(8):947-52. doi: 10.1038/sj.ejhg.5201428. PMID 15870827
- [Background] Derks TG, Reijngoud DJ, Waterham HR, Gerver WJ, van den Berg MP, Sauer PJ, Smit GP. The natural history of medium-chain acyl CoA dehydrogenase deficiency in the Netherlands: clinical presentation and outcome. J Pediatr. 2006 May;148(5):665-670. doi: 10.1016/j.jpeds.2005.12.028. PMID 16737882
- [Background] Derks TG, Boer TS, van Assen A, Bos T, Ruiter J, Waterham HR, Niezen-Koning KE, Wanders RJ, Rondeel JM, Loeber JG, Ten Kate LP, Smit GP, Reijngoud DJ. Neonatal screening for medium-chain acyl-CoA dehydrogenase (MCAD) deficiency in The Netherlands: the importance of enzyme analysis to ascertain true MCAD deficiency. J Inherit Metab Dis. 2008 Feb;31(1):88-96. doi: 10.1007/s10545-007-0492-3. Epub 2008 Jan 14. PMID 18188679
- [Background] Lamers KJ, Doesburg WH, Gabreels FJ, Lemmens WA, Romsom AC, Wevers RA, Renier WO. The concentration of blood components related to fuel metabolism during prolonged fasting in children. Clin Chim Acta. 1985 Oct 31;152(1-2):155-63. doi: 10.1016/0009-8981(85)90186-x. PMID 4053396
- [Background] Chang IJ, Lam C, Vockley J. Medium-Chain Acyl-Coenzyme A Dehydrogenase Deficiency. 2000 Apr 20 [updated 2024 Sep 26]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1424/ PMID 20301597
- [Background] Touw CM, Smit GP, Niezen-Koning KE, Bosgraaf-de Boer C, Gerding A, Reijngoud DJ, Derks TG. In vitro and in vivo consequences of variant medium-chain acyl-CoA dehydrogenase genotypes. Orphanet J Rare Dis. 2013 Mar 20;8:43. doi: 10.1186/1750-1172-8-43. PMID 23509891
- [Background] van der Hilst CS, Derks TG, Reijngoud DJ, Smit GP, TenVergert EM. Cost-effectiveness of neonatal screening for medium chain acyl-CoA dehydrogenase deficiency: the homogeneous population of The Netherlands. J Pediatr. 2007 Aug;151(2):115-20, 120.e1-3. doi: 10.1016/j.jpeds.2007.03.013. PMID 17643759
- [Background] van Veen MR, van Hasselt PM, de Sain-van der Velden MG, Verhoeven N, Hofstede FC, de Koning TJ, Visser G. Metabolic profiles in children during fasting. Pediatrics. 2011 Apr;127(4):e1021-7. doi: 10.1542/peds.2010-1706. Epub 2011 Mar 21. PMID 21422093